CLINICAL TRIAL: NCT02793570
Title: Native High-resolution 3D SSFP MR Angiography for Assessment of the Thoracic Aorta in Pregnant Subjects With Familial Aortopathies
Brief Title: Non-contrast 3D MR Angiography for Assessment of the Thoracic Aorta in Pregnancy
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, William E Moody, SpR Cardiology, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Magnetic Resonance Imaging; Pregnancy
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational

SUMMARY:
Introduction: Native magnetic resonance angiography (MRA) is recommended to assess the thoracic aorta during pregnancy, avoiding the risks of ionising radiation and contrast agent administration. This guidance is however, based only on consensus opinion supported by limited case reports (level of evidence C).

Aim: To evaluate the feasibility of performing native 3D steady-state free-precession (SSFP) MRA in pregnant subjects with inherited aortopathy to guide timing and mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant subject with a history of familial aortopathy

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant subjects in mid-trimester with familial aortopathy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Gestation at delivery | 40 weeks
Completion of non-contrast 3D MRA aorta | 40 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- QEHB, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://heart.bmj.com/content/102/Suppl_3/A13.abstract?sid=5d05d86c-f7e2-4c65-ad12-7b6e2c3b82f3